CLINICAL TRIAL: NCT01061476
Title: Sleep Apnea Treatment With Expiratory Resistance(Provent™)
Acronym: SATER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: ResMed (Industry); Ventus Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Susheel Patil, Assistant Professor of Medicine, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NA_00031257
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: sleep apnea; treatment; collapsibility; expiratory nasal resistance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm - Sleep apnea (Other): Participants with sleep apnea will be recruited for the study. Each participant will undergo 3 sleep studies to assess the effect of the Provent™ device. Participants will only use the device while they are in the sleep laboratory. They will not use the device at home between sleep studies .
  1. Baseline sleep study (No device) - Assess the effects of no Provent™ on sleep apnea severity.
  2. Treatment sleep study (Provent™ device used) - Assess the effects of Provent™ on sleep apnea severity
  3. Physiology sleep study (Provent™ on/off) - Assess the physiological effects of the Provent™ device on breathing during sleep.
  Interventions: Device: Treatment sleep study (Provent™ device used); Other: Baseline sleep study (No device); Other: Physiology sleep study (Provent™ on/off)

INTERVENTIONS:
Device: Treatment sleep study (Provent™ device used) — The patient's sleep apnea severity is determined on this night while using the Provent™ device. The patient only uses the Provent™ device on this night (single night use only).
Other: Baseline sleep study (No device) — The patient sleeps for 1 night in the sleep lab to determine their baseline sleep apnea severity without sleeping with the Provent device.
Other: Physiology sleep study (Provent™ on/off) — During this sleep study night, the patient is sleeping with a modified Provent™ device that can be turned on and off to assess changes in airflow during the night (single night use only).Provent™ on/off is bracketed in 10 minute intervals during stable stage 2 sleep.

SUMMARY:
Continuous positive airway pressure (CPAP) continues to be the primary therapy prescribed for the treatment of obstructive sleep apnea (OSA). Although effective, adherence to CPAP is suboptimal in many patients, making alternative therapies desirable. Recently, a novel device (Provent™) has been developed for the treatment of snoring and OSA. The purpose of the current study is to examine how well the Provent™ device treats OSA with particular attention to the how the it may treat sleep apnea and who may most likely benefit from the use of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults over the age of 18
* Diagnosed obstructive sleep apnea (defined as an RDI > 5 events per hour & ≥ 90% of disordered breathing events classified as obstructive)

Exclusion Criteria:

* Total sleep time from previous sleep study < 4 hours (240 minutes)
* Severe bilateral nasal obstruction (apparent mouth breathing at rest)
* Documented history of lung diseases, as defined below:
* Daytime hypercapnia (PaCO2 > 45 mmHg)
* Baseline SaO2 ≤ 92%
* Chronic lung disease except mild intermittent or mild persistent asthma
* Cor pulmonale
* Documented clinical cardiovascular disease, as defined below:
* Myocardial infarction in past 3 months
* Revascularization procedure in past 3 months
* Implanted cardiac pacemaker or ICD
* Unstable arrhythmias
* Congestive heart failure with ejection fraction < 40%
* Uncontrolled hypertension (BP > 190/110)
* History of end stage renal disease (on dialysis)
* History of end stage liver disease, such as:
* Jaundice
* Ascites
* History of recurrent gastrointestinal bleeding
* Transjugular intrahepatic portosystemic shunt (TIPS) ;
* Sleep disorders other than obstructive sleep apnea, such as:
* Narcolepsy
* Restless leg syndrome
* Periodic limb movements causing an arousal index of > 5 per hour
* Transportation industry worker (commercial truck or bus drivers, airline pilots)
* Known pregnancy (by self report)
* Known coagulopathy or anticoagulant use (e.g. coumadin) other than aspirin.
* Allergy to lidocaine

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susheel Patil, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Colrain IM, Brooks S, Black J. A pilot evaluation of a nasal expiratory resistance device for the treatment of obstructive sleep apnea. J Clin Sleep Med. 2008 Oct 15;4(5):426-33. PMID 18853699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 2010 and 2011. Patients were primarily recruited from the JH Sleep Disorders Center with a NREM RDI >= 10/h and >=90% of events were considered obstructive. 17 subjects met eligibility criteria with 12 enrolled.
Pre-assignment Details: Subjects were brought in for an evaluation prior to study enrollment to see if they would tolerate the Provent device by lying down with the device in place for 15-20 minutes.
Groups:
- Single Arm - Sleep Apnea: All participants will undergo 3 sleep studies - one off treatment, one on treatment, and one night to assess the physiological effects of the device on breathing during sleep.
  Provent™ : Provent™ is an expiratory nasal resistance device applied to the nares via adhesive.
Period: Overall Study
Arm/Group | Single Arm - Sleep Apnea
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm - Sleep Apnea
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in AHI
Description: The primary outcome was the change in the apnea hypopnea index (AHI). Sleep apnea events are defined as apneas and hypopneas.The AHI is a measure of sleep apnea severity. An AHI > 5 event/h is considered abnormal. AHI values are typically categorized as 5-15 events/hr = mild; 15-30 events/hr = moderate; and > 30 events/hr = severe. For this study we compared the change in AHI from the baseline sleep study (No Provent) compared to the treatment night sleep study (on Provent).
Time Frame: Comparisons were made between the 2 nights
Population: Although all participants went through the sleep studies, there was insufficient data in 1 subject to assess sleep apnea severity and was therefore excluded from analysis.
Measure: Mean (Standard Deviation); unit: events/h
Groups:
- Single Arm - Sleep Apnea: Each participant had 3 sleep studies. Sleep Study #1 - the patient did not have the Provent™ device on to assess baseline sleep apnea severity. On sleep study #2 - the patient used the Provent™ device to re-assess changes in sleep apnea severity. On sleep study #3, the patient used Provent™ for assessment of the physiological effects of the device on breathing during sleep.
  Participants did not use Provent™ outside of the sleep laboratory.
  Provent™ : Provent™ is an expiratory nasal resistance device applied to the nares via adhesive.
Arm/Group | Single Arm - Sleep Apnea
Number analyzed (Participants) | 11
events/h
  Baseline AHI | 45 (38)
  Change in AHI | -15.8 (18.02)

ADVERSE EVENTS:
Arm/Group | Single Arm - Sleep Apnea
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
* Small sample size and limited power for analysis.
* Oral breathing during expiratory nasal resistance (ENR) confounds the mechanism of action.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less